CLINICAL TRIAL: NCT04361227
Title: Prospective Study of Utility of OverStitch Sx Endoscopic Suturing System After ESD Procedure
Brief Title: Utility of OverStitch Sx After ESD
Status: Completed | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Mohamed Othman, Principal Investigator, Baylor College of Medicine
Other Study IDs: H-47184
Record Dates: First submitted 2020-04-22; First posted 2020-04-24 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Gastrointestinal Neoplasms
Keywords: Gastrointestinal Neoplasms; OverStitch Sx; Endoscopic Submucosal Dissection
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 48 Months
Biospecimen Retention: Samples With DNA — Gastrointestinal lesion/biopsy for pathological evaluation
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study is a prospective study where the investigators will make a database of all the patients who have received this procedure and will document various outcomes (i.e. number of sutures used, number of clips (if used), time required to close, complications/ issues). No changes will be done to the participant's procedure and the participants are asked to consent for the use of the participant's data in our database. The participants are being asked to be in this research study because the participants have been scheduled to undergo an ESD procedure at Baylor St. Luke Medical Center and will most likely require clipping and/or suturing following intervention. This study is important because this is a relatively new procedure; although it is a part of the participant's standard of care, it is not done in many hospitals. The investigators would like to document the outcomes and results of such procedures to continuously improve our standard of care.

DETAILED DESCRIPTION:
Resection of gastrointestinal neoplastic lesions at an early stage has been associated with improved clinical outcomes. While surgery has been traditionally performed for the resection of these precancerous or cancerous lesions confined to the mucosa of the GI tract, it is often associated with a higher morbidity and mortality rate compared to alternative endoscopic therapies. Recently, endoscopic submucosal dissection (ESD) has emerged as a new endoscopic technique that allows en-bloc resection of GI lesions, irrespective of size. In comparison to other endoscopic techniques, such as endoscopic mucosal resection (EMR), ESD is associated with higher curative resection rates and lower recurrence. While ESD was initially developed for the treatment of gastric cancer in Asia, which is relatively rare in the West, this technique would intuitively seem suitable for the resection of other superficial neoplastic lesions in the GI tract (i.e. large colon polyps, Barrett's mucosa, early non-invasive cancer). With the differences in patient population and disease location one can anticipate some differences in outcomes between ESD performed in Asian and US patients. Endoscopic Submucosal Dissection (ESD) is considered the gold standard for removal of pre-cancerous lesions from the GI tract, as histological analysis is more definitive, and the recurrence rate is lower as compared to endoscopic mucosal resection (EMR).

While ESD is useful for therapeutic and diagnostic purposes, the technique is rather difficult and detailed requiring extended procedure times. The most common complications of the ESD techniques are bleeding and perforation. Other rare complications include aspiration pneumonia, air embolisms, or stenosis. For this reason, closure of the mucosa following an endoscopic resection became an area of increased interest.

A randomized study in October of 2019 examined if prophylactic closure of a mucosal defect with clips would reduce the risk of bleeding following endoscopic intervention by EMR. 919 patients were randomly assigned to groups with 3.5% of patients experiencing post-procedure bleeding compared to 7.1% within the control group. Through this randomized trial, they found a significant reduction in post-procedural bleeding when patients undergo endoscopic clip closure of the mucosal defect.

With the advancements in endoscopic therapy, post-procedural clipping is now a well-established means of treatment following mucosal resections. Clipping, however, has two limitations including their inability to close large defects and the increasing difficulty in removal of those clips. To address these issues, endoscopic suturing systems have been developed which simulate the effectiveness of surgical stitching. The OverStitch Sx (Apollo Endosurgery Inc.) is commercially available and widely used in various applications such as the fixation of esophageal stents, suturing of ulcers, or reduction of anastamoses in bariatric surgeries.

Kantsevoy et al. in a 2014 retrospective study has shown that large mucosal defects treated with endoscopic suturing following an ESD resulted in a decrease rate of adverse events as well as the need for hospitalizations. All patient lesions were successfully and completely closed with no delayed or immediate adverse events following the procedure. The study concludes that the use of the Overstitch Sx device is fast and feasible and can decrease treatment costs by reducing the need to hospitalize patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18-99, who are scheduled to undergo ESD procedure with possible mucosal defect closure.

Exclusion Criteria:

* Age is less than 18 years old

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to/scheduled for ESD procedure at Baylor College of Medicine with possible mucosal defect closure.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2020-07-02 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
Clinical/technical success rate utilizing endosuture | 2 years
  To assess feasibility and technical success of using Overstitch Sx system for closure after ESD
Rate of patients reported with bleeding/perforation post-ESD procedure | 2 years
  Conduct follow-ups for risk of bleeding and perforation after closure
Closure time after ESD | 2 years
  Record time needed to close lesion

SECONDARY OUTCOMES:
Additional clip closure | 2 years
  Identify, if any, need for additional clipping after endoscopic suture closure
Clips used post-ESD | 2 years
  Record number of sutures needed to close lesion

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
Study is currently considered as a single-center prospective study.

REFERENCES:
- [Derived] Keihanian T, Zabad N, Khalaf M, Abdel-Jaber W, Kim YI, Jawaid SA, Abidi WM, Marginean EC, Othman MO. Safety and efficacy of a novel suturing device for closure of large defects after endoscopic submucosal dissection (with video). Gastrointest Endosc. 2023 Sep;98(3):381-391. doi: 10.1016/j.gie.2023.04.006. Epub 2023 Apr 14. PMID 37061137